CLINICAL TRIAL: NCT03040427
Title: The Role of F-18 Florbetapir in the Early Detection of Cardiac Amyloidosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: The Cleveland Clinic (Other)
Collaborators: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-960
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Amyloidosis
Keywords: F-18 florbetapir; Amyvid; PET scan; Early detection
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AL or TTR type amyloidosis (Experimental): The participants will undergo F-18 florbetapir PET scan.
  Interventions: Drug: F-18 florbetapir

INTERVENTIONS:
Drug: F-18 florbetapir — Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid).
  Other Names: Amyvid; Florbetapir-fluorine-18; 18F-AV-45

SUMMARY:
The investigators postulate that F-18 florbetapir will show improved detection of cardiac amyloidosis over conventional non-invasive imaging techniques, particularly in early disease.

DETAILED DESCRIPTION:
F-18 florbetapir is currently used for the early detection of brain amyloid (Alzheimer's disease). The hypothesis is that F-18 florbetapir will detect amyloid deposition in myocardium prior to current non-invasive diagnostic measures, particular electrocardiography with strain and technetium pyrophosphate scintigraphy. The investigators intend to use F-18 florbetapir and assess its correlation between standard non-invasive diagnostic modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with extra-cardiac biopsy-proven AL or ATTR amyloidosis
2. Patients with a ratio of affected to unaffected free light chains >5 or free light chain difference of >50

Exclusion Criteria:

1. Echocardiographic evidence of cardiac amyloidosis with septal and posterior wall thickness ≥ 13mm
2. Contraindication to florbetapir or its components
3. Refusal to participate in the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Nissen, MD, Study Chair — The Cleveland Clinic; Wael Jaber, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation (Main Campus), Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- At Risk for Symptomatic AL Cardiac Amyloidosis: Patients with MGUS at risk for developing AL amyloidosis
- At Risk for Symptomatic ATTR Cardiac Amyloidosis: Patients with biopsy proven extra-cardiac ATTR amyloidosis
- Control Patients: Negative carpal tunnel biopsy
Period: Overall Study
Arm/Group | At Risk for Symptomatic AL Cardiac Amyloidosis | At Risk for Symptomatic ATTR Cardiac Amyloidosis | Control Patients
Started | 2 | 6 | 4
Completed | 2 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | At Risk for Symptomatic AL Cardiac Amyloidosis | At Risk for Symptomatic ATTR Cardiac Amyloidosis | Control Patients | Total
Number analyzed (Participants) | 2 | 6 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (3.5) | 71.4 (5.2) | 72 (6.9) | 72 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 5 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Myocardial F18-florbetapir Uptake
Description: Number of participants with quantitative F18-florbetapir uptake above previously defined control values
Time Frame: at the time of the PET scan
Population: All participants had quantitative uptake of F18-Flobetapir
Measure: Count of Participants; unit: Participants
Arm/Group | At Risk for Symptomatic AL Cardiac Amyloidosis | At Risk for Symptomatic ATTR Cardiac Amyloidosis | Control Patients
Number analyzed (Participants) | 2 | 6 | 4
Participants | 2 | 6 | 4

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | At Risk for Symptomatic AL Cardiac Amyloidosis | At Risk for Symptomatic ATTR Cardiac Amyloidosis | Control Patients
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03040427/Prot_SAP_000.pdf